CLINICAL TRIAL: NCT02968784
Title: Focal ExAblate™ MR-Guided Focused Ultrasound (MRgFUS) Treatment for Management of Organ-Confined Intermediate Risk Prostate Cancer (OC-IRPC): Evaluation of Safety and Effectiveness
Brief Title: Focal ExAblate MR-Guided Focused Ultrasound Treatment for Management of Organ-Confined Intermediate Risk Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCa006
Record Dates: First submitted 2016-09-29; First posted 2016-11-21 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRgFUS; ExAblate; Focused Ultrasound
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate MRgFUS (Experimental): Up to 50% of the prostate gland will be treated. Treatment will include the Index lesion which is visible on MRI + tumor free margins of 3-mm; tumor free margins will not extend beyond the posterior aspect of the prostate capsule.
  Urethral and bilateral neurovascular bundle preservation will be preferred whenever clinically justified.
  Additional foci in the same hemisphere that are confirmed by biopsy and are < Gleason Score 7 (up to 3+4 or 4+3) or suspected to be positive for malignancy based on multi parametric-MRI) will also be included in the treated volume, providing total treatment volume does not exceed 50% of the gland.
  Interventions: Device: ExAblate MRgFUS

INTERVENTIONS:
Device: ExAblate MRgFUS — ExAblate treatment of prostate cancer less than or equal to Grade 7
  Other Names: Focused Ultrasound

SUMMARY:
This study is intended to show that ExAblate™ MRgFUS is a safe procedure that can significantly postpone or eliminate the need of patients with organ confined intermediate risk prostate cancer to undergo a definitive treatment (i.e., Radical Prostatectomy or Radiation therapy) for their disease.

DETAILED DESCRIPTION:
This study will evaluate the proportion of patients with organ-confined intermediate risk prostate cancer (OC-IRPC) undergoing focal ExAblate™ MRgFUS prostate treatment that will be free of clinically significant PCa which requires definitive treatment at 2 years after completion of their ExAblate™ treatment and to demonstrate the safety of focal ExAblate™ MRgFUS treatment.

Clinically significant PCa requiring definitive treatment is defined as pathology findings from whole-gland, imaging-guided, extended mapping biopsy of Gleason Score (GS) > 7

The primary efficacy endpoint in this trial, measured at 24 months with whole-gland extended imaging-guided mapping biopsy, is Response scored dichotomously for each subject as follows:

* Response = 0 ("Failure"): Positive mapping biopsy defined as Gleason Score > 7 (indicating definitive treatment) in any part of their prostate gland
* Response = 1 ("Success"): Negative mapping biopsy defined as Gleason Score < 7.

Safety of ExAblate™ treatment will be determined by evaluation of the incidence and severity of device related complications from the first treatment day visit throughout entire follow-up duration.

All adverse events will be captured and recorded. However, the safety of the ExAblate™ treatment will be defined by the incidence and severity of treatment or device related adverse events, grades III - V (CTCAE version 4.03; 2010-06-14).

Secondary Effectiveness Outcomes:

1. % of patients with negative 5-month follow-up biopsy results in the treated part of the prostate
2. Treatment effect on patients' Quality of Life (QoL), the following validated self-reported urogenital functioning assessment instruments will be used before and following treatment at pre-specified intervals.

   1. Urinary symptoms - IPSS
   2. Urinary continence - ICIQ-UI-SF
   3. Sexual function - IIEF-15
3. PSA levels and post-treatment PSA kinetics will also be assessed

ELIGIBILITY:
Inclusion Criteria:

* PSA ≤ 20 ng/ml
* Histologically proven PCa on imaging-guided transrectal or transperineal extended mapping biopsy
* Patient with intermediate risk, early-stage organ-confined prostate cancer (T1a up to T2b, N0, M0) and voluntarily chooses ExAblate thermal ablation as the non-invasive treatment, who may currently be on wtachful waiting or active surveillance and not in need of imminent therapy
* Gleason Score 7 (3+4 or 4+3) based on mapping prostate biopsy with no more than 15mm cancer in maximal linear dimension in any single core
* Single hemilateral index Gleason 7 lesion identified in the prostate based on biopsy mapping with supporting MRI findings; may have secondary Gleason 6 lesion on ipisilateral or contralateral side confirmed with biopsy and/or MRI

Exclusion Criteria:

* Any Contraindication to MRI, such as: over-size limitations avoiding patient's positioning in the bore of MRI scanner, claustrophobia, implanted ferromagnetic materials or foreign objects, or known contraindication to utilization of MRI contrast agent (e.g., Gadolinium/Magnevist)
* History of prostatectomy, radiation therapy to the pelvis for any other malignancy, brachytherapy, Cryotherapy, US-guided HIFU, orchiectomy, prostate photodynamic therapy, or prostate cancer-specific chemotherapy
* Patient under androgen deprivation therapy (ADT), alpha reductase inhibitors, and/or other hormonal treatment within the past 6 months
* Any rectal disease, pathology, anomaly, injury, previous treatment, or scarring which could change acoustic properties of the rectal wall, or might prevent safe probe insertion (e.g., inflammatory bowel disease, fistula, stenosis, fibrosis, or symptomatic hemorrhoids
* History of an invasive malignancy other than basal or squamous skin cancers in the last 5 years
* Existing urethral or bladder neck contracture/stricture
* Prostatitis NIH categories I, II and III
* Implant near (<1cm) the prostate

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-06; Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint in this trial measured with whole-gland extended imaging-guided mapping biopsy, is Response scored dichotomously; success vs. failure | 24 months post treatment
  Response will be based on mapping biopsy defined by Gleason 7 Score in any part of the prostate gland
Adverse events | 24 months post treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Percent of patients with negative biopsy | 5 months post treatment
  % of patients with negative 5-month follow-up biopsy results in the treated part of the prostate
Quality of Life - urinary symptoms - IPSS questionnaire score | 24 months post treatment
  Treatment effect on patients' Quality of Life (QoL), i.e., urinary symptoms
Quality of Life - urinary continence - ICIQ-SF questionnaire score | 24 months post treatment
  Treatment effect on patients' Quality of Life, (QoL), i.e., urinary continence
Quality of Life - sexual function - IIEF-15 questionnaire score | 24 months
  Treatment effect on patients' Quality of Life, (QoL), i.e.,sexual function
Prostate Specific Antigen (PSA) | 24 months post treatment
  PSA levels and post-treatment PSA kinetics will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sangeet Ghai, MD, Principal Investigator — Toronto General Hospital
Locations (4):
- Toronto General Hospital, Toronto, Ontario, Canada
- China (2):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
- St. Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided